CLINICAL TRIAL: NCT02404298
Title: Identification of the Mechanisms of Action of Intravenous Immunoglobulins in CIDP by Analysis of the Genetic Expression Profile in Blood Mononuclear Cells
Brief Title: Transcriptome Analysis of the Peripheral Blood in CIDP
Acronym: PHARMACOPID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P111122
Record Dates: First submitted 2015-02-06; First posted 2015-03-31 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Chronic Inflammatory Demyelinating Polyradiculoneuropathy; Autoimmune Diseases; Clarkson Syndrome; Muscular Autoimmune Disorders
Keywords: Transcriptome analysis; peripheral blood; chronic inflammatory demyelinating polyradiculoneuropathy; auto immune diseases; IVIg
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Autoimmune Diseases | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IVIg (Experimental)
  Interventions: Drug: IVIg

INTERVENTIONS:
Drug: IVIg

SUMMARY:
Chronic inflammatory demyelinating polyradiculoneuropathy (CIDP) is an immune-mediated disorder of peripheral nerves. Intravenous immunoglobulins (IVIg) are a first line therapy for CIDP. The investigators used a transcriptomic approach to compare the gene expression profiles in the peripheral blood of patients having a CIDP or autoimmune diseases, before and after IVIg treatment, in order to identify their mechanism of action in this condition, to lead to a better understanding of CIDP pathophysiology, and potentially determine factors associated with the response to the treatment.

DETAILED DESCRIPTION:
We study the change of the:

* gene profile on transcriptome analysis of peripheral blood
* T cell repertory
* igG dosage
* immunological profile

Before IVIG (T1 time) and and 3 weeks after IVIg treatment (T2 time). On a population of patients having: CIDP, autoimmune muscular disease, Clarkson syndrome, or autoimmune diseases.

We also search for polymorphism of FCgammareceptor, TKPC et CASP3 genes in CIDP patients

ELIGIBILITY:
Inclusion criteria :

* Age ≥ 18 years old
* Obtained informed consent
* Patient having a definite or probable CIDP according to EFNS/PNS criteria or atypical CIDP corresponding to patients having the EFNS/PNS clinical criteria and at least two EFNS/PNS supportive criteria
* Or
* Patient having a muscular autoimmune disease, or a Clarkson syndrome or other autoimmune disease
* Currently treated by IVIG

Exclusion criteria :

* pregnancy
* breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-02 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Gene expression profile | 3 weeks
  Change of the gene expression profile of a peripheral blood sample collected. just before IVIg administration (T1), and 3 weeks after IVIg treatment (T2)

SECONDARY OUTCOMES:
Gene expression profile in each lymphocytary sub-group | 3 weeks
  Change of the gene expression profile of a peripheral blood sample collected. just before IVIg administration (T1), and 3 weeks after IVIg treatment (T2), in each lymphocytary sub-group : CD3+CD4+, CD3+CD8+, CD4+FoxP3+, CD4+CD25+
IgG | 3 weeks
  To measure IgG in a peripheral blood sample at T1 and T2 time

CONTACTS AND LOCATIONS:
Overall Officials: Karine Viala, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Grooupe Hospitalier Pitié Salpetrière, Paris, France